CLINICAL TRIAL: NCT06087172
Title: Validity and Reliability of 6 Minutes Stepper Test in Hypertensive Patients
Brief Title: Validity of 6 Minutes Stepper Test in Hypertension
Status: Completed | Type: Observational
Sponsor: Ebru Calik Kutukcu (Other)
Responsible Party: Sponsor-Investigator, Ebru Calik Kutukcu, Associate Professor, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: GO 22/388
Record Dates: First submitted 2023-09-17; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Arterial Hypertension; Hypertension
Keywords: Stepper Test; Exercise Capacity; Cardiac Rehabilitation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertensive Individuals: Patients diagnosed with arterial hypertension
  Interventions: Diagnostic Test: Six Minutes Stepper Test (6MST)

INTERVENTIONS:
Diagnostic Test: Six Minutes Stepper Test (6MST) — Patients were applied two 6MST and 6MWT. 6MWT was conducted to test convergent validity of 6MST.
  Other Names: Six Minutes Walking Test (6MWD)

SUMMARY:
The six minutes stepper test (6MST) was used assess exercise capacity of individuals having different chronic conditions. In the literature, there are some validation studies analyzing validity of 6MST. In this study, the main aim was to analyse validation of 6MST in hypertensive individuals.

DETAILED DESCRIPTION:
6MST is a space-safe, feasible and sensitive test to assess exercise capacity. In the literature, there are lots of field tests assessing exercise capacity of individuals with chronic status. But common field tests eg 6MWT requires long spaces and it could become an important barrier in clinical settings. Hypertension is a common chronic disease and hypertensive individuals are important candidates of cardiac rehabilitation. As an important outcome assesing exercise capacity are very important before and after cardiac rehabilitation. In this study, the main aim was to investigate reliability and validity of 6MST in systemic hypertension.

ELIGIBILITY:
Inclusion Criterias:

* Being 18 to 65 years,
* Diagnosed with hypertension and willing to participate the study.

Exclusion Criterias:

* having a neurological, cognitive and/or orthopedic disease that affect the measurements,
* severe respiratory disease (FEV1 < 35%; FVC < 50%),
* presence of acute infection,
* any malignancy,
* dementia,
* any cardiovascular event in the last 6 months,
* uncontrolled hypertension and diabetes
* body mass index (BMI) higher than 40 kg/m2

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diagnosed with systemic (arterial) hypertension and convenient with inclusion and exclusion criterias.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
exercise capacity | through study completion two day
  steps during 6MST
functional capacity | through study completion two day
  walking distance during 6MWT

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, PhD, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)